CLINICAL TRIAL: NCT01322802
Title: A Phase I Trial of the Safety and Immunogenicity of a DNA Plasmid Based Vaccine Encoding the Amino Acids 1-163 of Insulin-Like Growth Factor Binding Protein-2 (IGFBP-2) in Patients With Advanced Ovarian Cancer
Brief Title: Vaccine Therapy in Treating Patients With Stage III-IV or Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7396; NCI-2011-00099 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 134; 7396 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); RG7212000 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2011-03-07; First posted 2011-03-25 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Stage III Ovarian Epithelial Cancer; Stage III Ovarian Germ Cell Tumor; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor
Keywords: Ovarian Cancer; Vaccine; Stage III; Stage IV; Remission
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (pUMVC3-hIGFBP-2 multi-epitope plasmid DNA vaccine) (Experimental): Patients receive pUMVC3-hIGFBP-2 multi-epitope plasmid DNA vaccine ID monthly for 3 months.
  Interventions: Biological: pUMVC3-hIGFBP-2 multi-epitope plasmid DNA vaccine; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: pUMVC3-hIGFBP-2 multi-epitope plasmid DNA vaccine — Given ID
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects of vaccine therapy in treating patients with stage III-IV or recurrent ovarian cancer. Vaccines made from deoxyribonucleic acid (DNA) may help the body build an effective immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of an insulin like growth factor binding protein 2 (IGFBP-2) Th polyepitope plasmid based vaccine in patients with advanced stage or recurrent ovarian cancer.

SECONDARY OBJECTIVES:

I. To determine the immunogenicity of IGFBP-2 Th polyepitope plasmid based vaccine in patients with advanced stage or recurrent ovarian cancer.

II. To determine whether intermolecular epitope spreading occurs with the generation of an IGFBP-2 specific Th1 immune response.

III. To determine whether IGFBP-2 vaccination modulates T regulatory cells.

OUTLINE:

Patients receive pUMVC3-hIGFBP-2 multi-epitope plasmid DNA vaccine intradermally (ID) monthly for 3 months.

After completion of study treatment, patients are followed up at 1, 3, 6, and 12 months, and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced stage (III/IV) or recurrent ovarian cancer who have been treated to complete remission with standard therapies including primary debulking surgery
* Cancer antigen 125 (CA-125) level within normal limits for the testing laboratory must be documented 90 days prior to enrollment when the assessment of CA-125 is applicable
* Patients must be at least 28 days post cytotoxic chemotherapy, and/or monoclonal antibody therapy, prior to enrollment
* Patients must be at least 28 days post systemic steroids prior to enrollment
* Patients must have Eastern Cooperative Oncology Group (ECOG) Performance Status Score of =< 2
* Patients must have recovered from major infections and/or surgical procedures, and in the opinion of the investigator, not have any significant active concurrent medical illnesses precluding protocol treatment
* Estimated life expectancy of more than 6 months
* White Blood Cell (WBC) >= 3000/mm^3
* Hemoglobin (Hgb) >= 10 mg/dl
* Hematocrit (Hct) >= 28%
* Serum creatinine =< 2.0 mg/dl or creatinine clearance > 60 ml/min
* Total bilirubin =< 2.5 mg/dl
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) =< 3 times upper limit of normal (ULN)
* Blood glucose < 1.5 ULN

Exclusion Criteria:

* Patients with any of the following cardiac conditions: symptomatic restrictive cardiomyopathy; unstable angina within 4 months prior to enrollment; New York Heart Association functional class III-IV heart failure on active treatment; symptomatic pericardial effusion
* Uncontrolled diabetes
* Patients with any contraindication to receiving sargramostim (rhuGM-CSF) based products
* Ovarian cancer of a low malignant potential phenotype or clear cell histology
* Patients with any clinically significant autoimmune disease uncontrolled with treatment
* Patients who are currently receiving an anti-IGF-IR monoclonal antibody as part of their treatment regimen
* Patients who are simultaneously enrolled in any other treatment study
* All subjects able to bear children

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03-06 (Actual); Primary Completion 2015-01-09 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Safety as assessed per Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 16 months
  Demographic and background characteristics obtained at enrollment will be listed and summarized. The type and grade of toxicities noted during the immunization regimen will be summarized. All adverse events noted by the investigator will be tabulated according to the affected body system. Descriptive statistics will be used to summarize changes from baseline in clinical laboratory parameters.

SECONDARY OUTCOMES:
Immunogenicity, via cellular immune response and humoral immune response, as assessed by the generation of IGFBP-2 specific T cells and IgG antibodies | Up to 16 months
  Cellular immune response will be defined by the magnitude of the Th1 antigen specific immune response using IFN-gamma enzyme-linked immunosorbent spot (ELISPOT). Humoral immune response will be measured by enzyme-linked immunosorbent assay (ELISA) and serum antibody avidity for IGFBP-2 using ELISA to determine an avidity index (AI) before and after vaccination. Spearman's correlation coefficient will be used to estimate the correlation between two continuous measures.
Epitope spreading with the generation of an IGFBP-2 Th1 immune response | Up to 16 months
  Peripheral blood mononuclear cells (PBMC) will be assessed by ELISPOT for immunity to a panel of immunogenic ovarian cancer related proteins: topoisomerase II-alpha (a), p53, IGF-IR, FASCIN-1, and MMP-7. Epitope spreading will have been considered to occur if new immune responses are generated to any of these antigens during the course of the study. In addition, epitope spreading and T regulatory cells will be defined as present or absent, and the probability of each will be estimated as a simple proportion as above with toxicity.
Levels of regulatory T- cells (Tregs) over the course of immunization to detect modulation of Tregs with vaccination | Up to 16 months
  Assessed by flow cytometry of PBMC. In addition, epitope spreading and T regulatory cells will be defined as present or absent, and the probability of each will be estimated as a simple proportion as above with toxicity.
Disease-free survival | Up to 5 years
  A questionnaire will be sent to the patient's primary oncologist requesting laboratory evaluation of toxicity, CA-125, and the patient's disease free and overall survival status.
Overall survival | Up to 5 years
  A questionnaire will be sent to the patient's primary oncologist requesting laboratory evaluation of toxicity, CA-125, and the patient's disease free and overall survival status

CONTACTS AND LOCATIONS:
Overall Officials: Mary Disis, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States